CLINICAL TRIAL: NCT01834833
Title: Consultation at 8 Days to Reduce Hospitalisations in Heart Failure Patient.
Acronym: CHIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P110601 - PHRQ1104
Record Dates: First submitted 2013-01-17; First posted 2013-04-18 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; rehospitalisation; education; follow-up

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): usual care without systematic cardiology evaluation between 1 and 2 weeks
- Follow-up (Experimental): Evaluation by a cardiologist using echocardiography, completed by education of the patient if necessary
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Evaluation by a cardiologist using echocardiography, completed by education of the patient if necessary
  Arms: Follow-up

SUMMARY:
Evaluate the benefit of systematic appointment with a cardiologist a week after hospitalisation for acute heart failure. Randomised, endpoint: number of day alive out of hospital during 6 months

DETAILED DESCRIPTION:
Background: the risk for rehospitalisation is very high after hospitalisation for acute heart failure. Aim: evaluate the benefit of a consultation with a cardiologist, including echocardiography and education of the patient, between 7 and 15 days after discharge, in high risk patients, identified with BNP or incomplete therapy. Parallel randomised study. The main endpoint is the number of day alive out of hospital during the 6 months post discharge; statistics intention to treat comparison of the number of days alive out of hospital in the group with consultation compared with the group without consultation. Recruitment 3 years and 4 months, follow-up 6 months. Patients included have been hospitalised in hospital BICHAT 75018 Paris, France. Financing is by the ministry of health (PHRQHOS)

ELIGIBILITY:
Criteria of inclusion :

* Patient with decompensated heart failure hospitalized in the hospital BICHAT,
* For whom is planned a return at home,
* Valid (being able to return for a consultation to the hospital)
* Having Nt-ProBNP of exit ≥ 3500 ng /l and/or a non optimized treatment of exit - according to the doctor who has it the responsibility,
* Having signed the consent form by participation in the study.

Criteria of not inclusion :

* Age < 18 years,
* Not membership in a national insurance scheme or in the Universal Health
* Coverage (CMU)(FREE UNIVERSAL HEALTH CARE)(A patient benefiting from the Medical aid of the State (AME) cannot be included)
* Participation to another protocol of research,
* Not being reachable by telephone in 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
days alive out of hospital 6 months post discharge | 6 months

SECONDARY OUTCOMES:
rehospitalisation rate at 6 months | 6 months
mortality at 3 and 6 months | 3 and 6 months
number of patients receiving beta-blocker at 6 months | 6 months
number of patients receiving a ACEI at 6 months | 6 months
QOL at 6 months | 6 months
autoevaluation of improvement/alteration of the patient state at 6 months | 6 months
number of patients receiving beta-blocker at 3 months | 3 months
number of patients receiving a ACEI at 3 months | 3 months
QOL at 3 months | 3 months
autoevaluation of improvement/alteration of the patient state at 3 months | 3 months
number of patients having an optimal treatment at 6 months | 6 months
number of patients having an optimal treatment at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume JONDEAU, MD, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Bichat Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided